CLINICAL TRIAL: NCT07080788
Title: Can Smoking Cessation Improve Physiological Markers of Chronic Pain Risk in Native American Smokers?: A Pilot Feasibility Study
Brief Title: Oklahoma Study of Native American Pain Risk IV: Smoking Cessation and Pain
Acronym: OK-SNAP IV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18695
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation Intervention; Pain; Smoking (Tobacco) Addiction
Keywords: Smoking cessation; Quantitative sensory testing
MeSH Terms: conditions — Pain; Smoking; Behavior, Addictive; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Smoking Cessation (Experimental)
  Interventions: Behavioral: Smoking Cessation

INTERVENTIONS:
Behavioral: Smoking Cessation — Investigators will provide financial incentives for biochemically verified abstinence at 4 weeks following treatment. This incentive is consistent with recent research using macro-level financial incentives and incorporates both short-term and long-term incentives to shape behavior.

SUMMARY:
The goal of this pilot study is to assess whether 4-weeks of verified smoking abstinence following financial incentive treatment for smoking cessation improves physiological markers of chronic pain risk in adult Native American smokers.

The main aims to answer are:

1. Determine study feasibility.
2. Obtain effect sizes for changes in pain amplification and pain inhibition in abstinent vs non-abstinent Native Americans.
3. Obtain effect sizes for variables in the conceptual model of the Native American smoking-pain relationship.

DETAILED DESCRIPTION:
Native Americans experience the highest rates of chronic pain of all U.S. racial/ethnic groups, and we have shown this disparity is partly explained by disrupted physiological pain regulation mechanisms, i.e., enhanced pain amplification and impaired pain inhibition. One unexplored variable that could disrupt these mechanisms in Native Americans is non-ceremonial tobacco smoking. Native Americans have the highest smoking rate in the U.S., and smoking is associated with disrupted pain regulation in non-Native American samples. Thus, there is a critical need to understand whether smoking contributes to NA pain risk.

There is high comorbidity between smoking and chronic pain, but it is also known that chronic pain patients who quit smoking have improved pain. This study aims to better understand the relationship between Native American smoking and chronic pain risk. It is believed that smoking increases chronic pain risk in pain-free Native Americans by increasing pain amplification and impairing pain inhibition, and smoking abstinence will reduce pain amplification and increase pain inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Native American/American Indian
* Currently smoking > 10 cigarettes per day but interested in quitting
* Own a smartphone with a data plan
* Ability to speak and read English

Exclusion Criteria:

* >18 years of age
* Currently pregnant
* Self-reported history of cardiovascular, neuroendocrine, musculoskeletal, or neurological disorders
* Current chronic pain
* Use of medication that could interfere with testing (e.g., recent use of analgesics, antidepressants, or anti-anxiety medications)
* Pepper allergy
* Inability to speak English
* Angina, arrhythmias, hypertension, heart disease
* Current psychosis (assessed by Psychosis Screening Questionnaire)
* Serious cognitive impairment (assessed by <20 score on the Montreal Cognitive Assessment [MoCA])

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pain inhibition | Baseline (1 day prior to smoking cessation treatment allocation) and Post-Treatment (following 4 weeks of treatment + 4 weeks of verified smoking abstinence)
  Pain inhibition will be assessed using a conditioned pain modulation task with cold water as the conditioning stimulus and electric stimulations as the test stimulus.
Inhibition of pain-related spinal reflex | Baseline (1 day prior to smoking cessation treatment allocation) and Post-Treatment (following 4 weeks of treatment + 4 weeks of verified smoking abstinence)
  Pain-related spinal reflex inhibition assessed from electromyogram will be assessed using a conditioned pain modulation task with cold water as the conditioning stimulus and electric stimulations as the test stimulus.
Allostatic load | Baseline (1 day prior to smoking cessation treatment allocation) and Post-Treatment (following 4 weeks of treatment + 4 weeks of verified smoking abstinence)
  A single latent variable for allostatic load will be created using principal components analysis to combine cardiovascular (i.e., resting blood pressure and heart rate and fasting lipid profile [HDL, LDL, total cholesterol, and triglycerides]), metabolic (i.e., BMI, waist-to-hip ratio, HbA1c), immune (i.e., hs-CRP), and parasympathetic (i.e., resting heart rate variability) variables.
Pain amplification | Baseline (1 day prior to smoking cessation treatment allocation) and Post-Treatment (following 4 weeks of treatment + 4 weeks of verified smoking abstinence)
  Pain amplification will be assessed by capsaicin (substance from hot chili peppers) pain model. Pain amplification is defined as the area of skin (in cm squared) surrounding the site of capsaicin application that shows higher pain relative to the untreated skin.

SECONDARY OUTCOMES:
Temporal summation of pain | Baseline (1 day prior to smoking cessation treatment allocation) and Post-Treatment (following 4 weeks of treatment + 4 weeks of verified smoking abstinence)
  Temporal summation of pain will be measured by assessing the change in a participant's pain ratings in response to identical noxious stimuli delivered in a rapid succession.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Rhudy, PhD, Principal Investigator — University of Oklahoma Health Sciences
Locations (1):
- University of Oklahoma - Schusterman Center, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and metadata will reside with the PI, research team, and tribal partners and made available to others following review, by the PI and tribal IRBs, of the data request. Requests for data will be made available as soon as possible, but no later than time of an associated publication. Those investigators approved to use data will be instructed to submit any products for tribal IRB review and approval before they are submitted for publication or presentation. If the goals of the approved request are outside the aims of the parent project, the requesting investigators may be required to reconsent participants before they are allowed access to data.
Time Frame: De-identified data will become available following publication of all findings (around 6/1/2030)
Access Criteria: To obtain access to the data, interested parties can contact the PI (jamie-rhudy@ouhsc.edu